CLINICAL TRIAL: NCT01148095
Title: A Single Centre Two Part Randomized Phase I Study to Assess the Pharmacokinetics of an ER Formulation of AZD2516 and to Assess the Safety, Tolerability and Pharmacokinetics of AZD2516 After Multiple Ascending Doses in Healthy Volunteers
Brief Title: To Investigate the Safety, Tolerability and Pharmacokinetics of AZD2516 After Multiple Dosing in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Quintiles, Inc. (Industry)
Responsible Party: MSD, AstraZeneca
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D2080C00002
Record Dates: First submitted 2010-06-18; First posted 2010-06-22 (Estimated); Last update posted 2011-02-08 (Estimated); Status verified 2011-02

CONDITIONS: Part A Healthy Young Males and Non-fertile Female Volunteers Aged 20 to 45 Years.; Part B Healthy Young Males and Non-fertile Female Volunteers Aged 20 to 45 and Elderly Volunteers Aged 60 to 80
Keywords: AZD2516; Phase 1; Healthy volunteer; pharmacokinetics; safety; tolerability; Multiple ascending doses

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): AZD2516 (dose escalating)
  Interventions: Drug: AZD2516
- 2 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AZD2516 — Oral, single, daily, 11 days
  Arms: 1
Drug: Placebo
  Arms: 2

SUMMARY:
AZD2516 is being developed for the oral treatment of chronic neuropathic pain. This study is split in to two parts. Part A will measure the effect of food and a new formulation of the drug in the blood and see how well it is tolerated. Part B will commence after the completion of Part A and will investigate the safety and tolerability of daily dosing with AZD2516.

ELIGIBILITY:
Inclusion Criteria:

* Have a body mass index (BMI) between 18 and 30 kg/m2 and weigh at least 50 kg and no more than 100 kg
* Healthy volunteers able and willing to comply with all study requirements.

Exclusion Criteria:

* An ongoing or history of a medical or psychiatric disease/condition which may put the healthy volunteer at risk or interfere with the study objectives because of participation in the study, as judged by the investigator(s).
* History of psychotic disorder among first degree relatives.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2010-06; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Adverse Events, vital signs | Day -1 until follow-up

SECONDARY OUTCOMES:
Maximum plasma concentration (Cmax) | Day 1 - Day 12
Time to Cmax (tmax) | Day 1 - Day 12
Terminal rate constant (λz) | Day 1 - Day 12

CONTACTS AND LOCATIONS:
Overall Officials: Darren Wilbraham, MBBS, DCPSA, Principal Investigator — Quintiles Drug Research Unit 6, Newcomen Street, London, SE1 1YR
Locations (1):
- Research Site, London, United Kingdom